CLINICAL TRIAL: NCT00175292
Title: A Randomized and Placebo-Controlled Double-Blind Multicentre Study to Determine the Efficacy and Safety of VSL#3 Probiotic Food Supplement Mixture in Prevention of Endoscopic Recurrence in Crohn's Disease Patients With Ileocolonic Surgical Resection and Small Intestine to Colon Anastomosis.
Brief Title: A Randomized Controlled Trial of VSL#3 for the Prevention of Endoscopic Recurrence Following Surgery for Crohn's Disease.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VSL-FED-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-05-14 (Estimated); Status verified 2008-05

CONDITIONS: Crohn's Disease; Inflammatory Bowel Disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

INTERVENTIONS:
Drug: Probiotic - VSL#3

SUMMARY:
This randomized placebo-controlled double-blind, multi-centre trial will determine the efficacy of the probiotic VSL#3 in the prevention of Crohn's disease development following surgical resection and re-anastomosis. A total of 120 patients will be randomly assigned in a 1:1 ratio to receive VSL#3 or placebo for 90 days. Patients who respond to study treatment, as defined by the absence of a severe endoscopic recurrence at day 90, will be offered open-label VSL#3 for an additional 9 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 16 years of age or older
2. Diagnosis of Crohn's disease
3. Resection of ileocolonic Crohn's disease and small bowel to colonic anastomosis within 30 days of randomization
4. Able to provide informed written consent
5. Women of child-bearing potential with a negative serum pregnancy test, and/or use of effective contraception

Exclusion Criteria:

1. Use of perioperative steroids in tapering doses and anti-diarrheal agents
2. Treatment with a TNF-antagonist in the 8 weeks prior to resection
3. Clinically significant Crohn's disease elsewhere in the GI tract
4. Clinically documented short bowel syndrome
5. Serious disease other than Crohn's disease
6. Impaired liver or renal function
7. History of cancer with less than 2 years disease-free state
8. Abnormal Laboratory values
9. Alcohol or drug abuse
10. Some psychiatric conditions
11. Patients using other study medications
12. Patients who are unable to attend study visits or comply with study procedures
13. Positive pregnancy test

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2003-12

PRIMARY OUTCOMES:
Prevention of severe endoscopic recurrence of Crohn's disease.

SECONDARY OUTCOMES:
Endoscopic recurrence at 90 days and 360 days
Crohn's Disease Activity Index (CDAI)
Quality of life
Safety and tolerance of VSL#3

CONTACTS AND LOCATIONS:
Overall Officials: Richard Fedorak, MD, Principal Investigator — University of Alberta
Locations (17):
- Canada (17):
  - Health Sciences Centre, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Walter Mackenzie Health Sciences Centre, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Dr. D.M. Petrunia, Inc., Victoria, British Columbia
  - Health Sciences Centre, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Surrey GI Clinic, Guelph, Ontario
  - McMaster University Medical Centre, Hamilton, Ontario
  - Hotel-Dieu Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Hopital St-Sacrement, Québec, Quebec

REFERENCES:
- [Derived] Fedorak RN, Feagan BG, Hotte N, Leddin D, Dieleman LA, Petrunia DM, Enns R, Bitton A, Chiba N, Pare P, Rostom A, Marshall J, Depew W, Bernstein CN, Panaccione R, Aumais G, Steinhart AH, Cockeram A, Bailey RJ, Gionchetti P, Wong C, Madsen K. The probiotic VSL#3 has anti-inflammatory effects and could reduce endoscopic recurrence after surgery for Crohn's disease. Clin Gastroenterol Hepatol. 2015 May;13(5):928-35.e2. doi: 10.1016/j.cgh.2014.10.031. Epub 2014 Nov 6. PMID 25460016